CLINICAL TRIAL: NCT03790202
Title: Open Label Assessment of VistaCare® Treatment in Current Medical Practice in Patients With Acute and Chronic Leg Wounds.
Brief Title: VistaCare® in the Treatment of Wounds of the Lower Extremity
Status: Completed | Type: Observational
Sponsor: DTAMedical SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: VistaCare® OPEN PMCF
Record Dates: First submitted 2018-12-24; First posted 2018-12-31 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Wound Heal
Keywords: wound; VistaCare; wound healing; controlled atmosphere
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- single cohort of up to 30 patients: patients with acute or chronic lower limb wounds to be treated with the VistaCare® device
  Interventions: Device: VistaCare®

INTERVENTIONS:
Device: VistaCare® — Controlled atmosphere wound healing device

SUMMARY:
Assessment of the safety and performance of the VistaCare® medical device in current medical practice in the treatment of acute and chronic lower limb wounds.

DETAILED DESCRIPTION:
The study is an open-label, prospective, multicenter, post-CE mark (European Conformity assessment indicating marketing approval in Europe) study to assess the safety and performance of the VistaCare® device in the treatment of wounds. The duration of patient follow-up is up to 30 days, with intermediate visits at 3, 7, 15 and 30 days following initiation of treatment with the device.

Up to 30 patients will be recruited in the trial. Assessments will include clinical status, wound status, standardized photography, TcPO2 (trans-cutaneous oxygen pressure assessment) in a study sub-population, visual analogy scales to assess pain and comfort and adverse events monitoring.

ELIGIBILITY:
Inclusion Criteria:

* male or female consenting and able patients aged 18 or more affiliated to social security
* presenting with acute or chronic traumatic or surgical lower limb wounds (excluding tumoral excision)
* presenting with no intercurrent pathology which in the opinion of the investigator may interfere with the capacity for wound healing
* patients whose wound is compatible in terms of location with VistaCare treatment
* patient whose wound has a minimal surface of 10 cm2
* patient whose wound does not need surgical Peterson after inclusion (if needed should be performed prior to inclusion)

Exclusion Criteria:

* Female patients pregnant, lactating, or of childbearing age and not using adequate contraception (pregnancy test mandatory)
* patients incapable of making an informed decision about participation
* patients presenting a condition that interferes with adequate wound healing capacity (uncontrolled diabetes, heavy smokers, auto-immune disease)
* concurrent treatment or treatment within one month prior to inclusion with local or systemic corticosteroids, immunosuppresseurs, chemotherapy or radiotherapy
* wound location incompatible with VistaCare
* general infection signs at the time of inclusion (fever, lymphangitis, pus ...)
* patients presenting with important uncontrolled hemorrhage at the time of inclusion
* patients previously recruited into this trial or any other trial within 1 month, or currently in the exclusion timeframe of another trial
* patients with a wound surface less than 10 cm2
* patient with a would previously treated with hyperbaric chamber
* legally incapacitated, under guardianship or psychiatric patients
* emergency condition prohibiting adequate patient consent prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients addressed to the hospital investigators, aged 18 and more, suffering from acute or chronic lower extremity wounds
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the global Safety of use of the VistaCare® medical device in standard medical practice | up to 30 days
  Assessment of the global safety of VistaCare® in current medical practice in patients with acute or chronic lower limb wounds through monitoring of concurrent averse events throughout the study duration. This will be assessed through the frequency of occurrence of device-related events, throughout the patient's participation in the trial
Assessment of the global Performance of the VistaCare® device in standard medical practice | up to 30 days
  Assessment of the global performance of the VistaCare® medical device as compared to its labeled performance in the approved indication (wound healing). This will be assessed through a global clinical assessment by the investigator of the wound improvement condition throughout the study visits, measured in 3 grades ranging from Aggravation (worst assessment), through Static (no improvement) to Improved (best assessment), taking into consideration the wound healing stage and general clinical condition per investigator's assessment.

SECONDARY OUTCOMES:
Assessment of time under VistaCare treatment till secondary treatment decision | up to 15 days
  Assessment of the time in days till decision to wound coverage, graft, wound dressing, or no further treatment needed and patient discharge. Duration in days from VistaCare treatment initiation to decision-making will be tabulated for each patient.
Wound surface calorimetric assessment of wound status | 30 days
  Description of wound clinical status evolution through photography, wound measurement in mm2 and visual assessment of wound status. This measure is based on the surface in mm2 of the wound components on a standard photography, each wound potentially comprising 3 wound stages surfaces : necrotic (worst), granulation and epithelization (most favorable wound healing stage). Those stages are measured on each visit on a standardized photography of the wound and the wound stage evolution in time is assessed for each patient by an external reviewer. Wound staging for each patient will be analyzed in time throughout patient's participation and presented as graphs.
Safety assessment of the VistaCare® treatment through monitoring of the frequency of adverse events | throughout 30 days
  Safety assessment of the VistaCare® treatment through adverse events monitoring, with frequency of patients presenting with any adverse event and frequency of each adverse event type, namely non-serious unrelated or device-related event (respectively AE, ADE), serious unrelated event (SAE), serious device-related event (SADE), unanticipated device-related event (UADE), or device deficiency. Tabulation of frequencies in percentages of patient occurrence and number of events per patient will be provided.
TcPO2 assessment | up to 30 days
  In a sub-group of up to 10 patients, measure of the trans-cutaneous oxygen pressure (TcPO2) around the wound to assess status and potential correlation with wound status. This measure is expressed in mmHG and the correlation between this measure and the wound healing stage will be statistically assessed to indicate if wound healing may be correlated to the oxygen pressure measure.
Quality of Life assessments | throughout 30 days
  Patient visual analogy scale (VAS) assessments of pain and comfort. Those scales are each graduated from 0 (none) to 10 (maximum pain or discomfort). The evolution in times of such scores will be statistically assessed for each patient.
Duration of hospitalization | throughout 30 days
  Assessment of the total duration of patient hospitalization in days.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Casanova, MD Pr, Principal Investigator — Hôpital de la Conception, Marseille, France; Regis Legré, MD Pr, Principal Investigator — Hôpital de la Timone, Marseille, France; Pierre-Edouard Magnan, MD Pr, Principal Investigator — Hôpital de la Timone, Marseille, France; Pascal Desgranges, MD Pr, Principal Investigator — CHU Henri Mondor, Créteil, France; Franck Duteille, MD Pr, Principal Investigator — CHU Nantes, France
Locations (4):
- France (4):
  - CHU Henri Mondor, Créteil
  - Hôpital La Timone, Marseille
  - Hôpital de la Conception, Marseille
  - CHU de Nantes Centre des Brûlés, Nantes

IPD SHARING:
Plan to Share IPD: No